CLINICAL TRIAL: NCT02775682
Title: Cerebral Autoregulation in Patients With Epilepsy
Acronym: CAPE
Status: Completed | Type: Observational
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Associated Dean of First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Other Study IDs: CA&EEG
Record Dates: First submitted 2016-05-13; First posted 2016-05-18 (Estimated); Last update posted 2021-08-25 (Actual); Status verified 2017-03

CONDITIONS: Epilepsy
Keywords: epilepsy, dynamic cerebral autoregulation
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- patients with epilepsy
- normal individuals without epilepsy

SUMMARY:
The purpose of this study is to determine whether patients with epilepsy exhibiting impaired dCA, which may contribute to subsequent stroke.

DETAILED DESCRIPTION:
The relationship between epileptic seizures and cerebrovascular disease is complex, ranging from mechanisms to clinical manifestation. Stroke is one of the most common causes of epilepsy in adulthood. It was also reported that patients with epilepsy exhibited a higher risk of stroke. But its potential mechanism was never fully understood. Dynamic cerebral autoregulation(dCA), a mechanism to maintain the cerebral bold flow, has been proved to be critical for the occurrence ,development and prognosis of ischemic neurovascular disease. In this study, we hypothesis that impaired dCA play a role in epilepsy and subsequent stroke.

ELIGIBILITY:
Inclusion Criteria:

* patients with epilepsy, as diagnosed by EEG

Exclusion Criteria:

* patients with status epilepticus
* intracranial and/or extracranial major vascular stenosis/occlusion diagnosed by a transcranial Doppler (EMS-9PB, Delica, China) and carotid ultrasound (IU22, Phillips, Andover, MA)
* a prior symptomatic cerebral vascular disease
* a history of hypertension, cardiovascular disease, diabetes, hyperlipemia, current arrhythmia, hyperthyroidism, anemia and unstable blood pressure, which may undermine hemodynamic stability, or inability to cooperate sufficiently to complete the cerebral auto regulation examination
* insufficient bilateral temporal bone windows for insonation of the middle cerebral artery
* intolerance to cerebral autoregulation measurements

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients with a diagnosis of epilepsy were recruited from the Department of Neurology, First Hospital of Jilin University, China. Patient was diagnosed with epilepsy by two neurologists according to the consequence of EEG.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
phase difference(PD) in degree | 1 year
  A dynamic cerebral auto-regulation parameter derived from transfer function analysis.Continuous cerebral blood flow velocities of bilateral middle cerebral artery will be assessed noninvasively using transcranial Doppler. Spontaneous arterial blood pressure will be simultaneously recorded using a servo-controlled plethysmograph on the left or right middle finger with an appropriate finger cuff size. Transfer function analysis will be used to derive the autoregulatory parameters.

SECONDARY OUTCOMES:
the rate of recovery of cerebral blood flow velocity | 1 year
  A dynamic cerebral auto-regulation parameter derived from transfer function analysis.The details are same as primary outcome
gain in cm/s/mmHg | 1 year
  A dynamic cerebral auto-regulation parameter derived from transfer function analysis.The details are same as primary outcome
the consequence of electroencephalograph（EEG） | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yi Yang, MD,PhD, Study Chair — Neuroscience Center, Department of Neurology, The First Hospital of Jilin University
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

REFERENCES:
- [Derived] Lv S, Guo ZN, Jin H, Sun X, Jia M, Ma H, Lv Y, Qiu Q, Liu J, Yang Y. Compromised Dynamic Cerebral Autoregulation in Patients with Epilepsy. Biomed Res Int. 2018 Feb 7;2018:6958476. doi: 10.1155/2018/6958476. eCollection 2018. PMID 29568762